CLINICAL TRIAL: NCT02429596
Title: A Randomized Controlled Trial of Generic Substitution of Antiepileptic Drugs
Brief Title: A Trial of Generic Substitution of Antiepileptic Drugs
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: FARM9A8J83
Record Dates: First submitted 2014-11-14; First posted 2015-04-29 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2015-04

CONDITIONS: Epilepsy
Keywords: antiepileptic drugs; generic substitution
MeSH Terms: conditions — Epilepsy | interventions — Lamotrigine; Levetiracetam; Topiramate; Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Experimental Treatment (Experimental): AED(s) currently taken (CBZ, VPA, TPM, OXC, LEV, LTG) will be substituted, starting with the morning dose on day 2, with an equivalent formulation available in the market. Namely, a brand product will be switched to a generic, randomly chosen among those available in the market, while maintaining unaltered the dosing regimen and times of administration.Likewise, a generic product will be switched to the brand or another generic.
  Interventions: Drug: Experimental
- No Experimental Treatment (No Intervention): When the randomized allocation requires continuation on the same product (control), the AED product(s) currently taken will be continued unaltered, with the same dosing regimen and times of administration.

INTERVENTIONS:
Drug: Experimental — Switch from brand to generic
  Other Names: Lamictal; Acido Valproico; Keppra; Topamax; Tegretol; Tolep
  Arms: Experimental Treatment

SUMMARY:
Background. Anecdotal reports and uncontrolled studies have described an association between generic substitution of antiepileptic drugs (AEDs) and adverse events, including loss of seizure control. Although these results are likely to be influenced by methodological bias, they have led to a strong opposition, among physicians and patients, to the use of generic products in epilepsy.

Objectives. The primary objective is to assess potential risks associated with substitution of the currently taken AED product with an equivalent product, using as endpoint changes in serum drug levels at steady-state after substitution compared with baseline. Secondary objectives will be the assessment of inter-subject variability in serum drug concentration on an unchanged treatment schedule, and evaluation of potential short-term changes in seizure control and adverse events rate.

Methods. The study will use an experimental randomized open-label non-inferiority design. The population will consist of 200 adults stabilized on chronic treatment with carbamazepine, valproic acid, topiramate, oxcarbazepine, levetiracetam or lamotrigine and admitted to hospital for diagnostic evaluation or other indications, with no expected treatment changes during the subsequent 5 to 6 days. Patients will be randomized to two groups. One group will continue to receive the AED products used before enrollment (brand or generic), whereas the other group will be switched to an alternative equivalent product. Dosing schedules of the AEDs being tested as well as comedications will be unaltered throughout the 6- to 7day period of the study. Serum AED levels (mean of two values obtained at peak and trough, respectively in the evening and the next morning) will be measured on day 1 (baseline) and 5 days post-randomization (6 days for patients receiving AEDs with half-lives above 12 h). The primary outcome endpoint will be the proportion of patients who, post-randomization, show a greater than 25% change in serum drug concentration compared with baseline. Secondary endpoints will include comparison of distributions of rough serum concentration changes between groups, other pharmacokinetic parameters, time to first seizure, total number of seizures, and adverse events.

DETAILED DESCRIPTION:
The primary objective is to provide high-quality evidence on potential risks associated with substitution of the currently taken AED product (carbamazepine,valproic acid, topiramate, oxcarbazepine, levetiracetam or lamotrigine) with an equivalent product, using as endpoint changes in serum drug levels at steady-state after substitution compared with baseline. Secondary objectives will be the assessment of inter-subject variability in serum drug concentration on an unchanged treatment schedule, and evaluation of potential short-term changes in seizure control and adverse events rate.

The study uses an experimental randomized non-inferiority design, and the hypothesis tested is that substitution of the currently taken AED product with another product (either generic or brand) will be associated with changes in serum drug levels which are no greater than those observed in a control group not undergoing any substitution.

The primary endpoint is the proportion of patients who post-randomization, will show a greater than 25% change in serum drug concentration compared with baseline.

The study will be conducted according to an experimental, prospective, randomized, open-label controlled, parallel-group design.

The study will be conducted in adults of either gender, enrolled at the time of hospital admission (or already hospitalized).

On the day of admission or inclusion in the study (day 1), all subjects fulfilling the eligibility criteria and enrolled in the study will be allocated by 1:1 randomization to two groups, using a centralized telephone-based randomization office located at the coordinating institution and stratification to ensure that the proportion of patients receiving a brand or a generic at baseline is comparable between groups. For subjects taking concomitantly more than one AEDs being tested, separate randomizations will be conducted separately for each AED (for example, a subject receiving valproic acid and carbamazepine will be randomized to continue on the same formulation of valproic or to switch to a different formulation of valproic acid, and at the same time separately randomized to continue on the same formulation of carbamazepine or to switch to a different formulation of carbamazepine).

On day 1 (day of admission or day of inclusion in the study), all subjects will continue to receive their current AED treatment, without any change in formulation (brand or specific generic product), route and dosing schedule. Two blood samples for the determination of the serum levels of the AED(s) will be collected, one on day 1 two hours after the evening dose (absorptive phase sample, close to the expected peak time) and one the next morning (day 2) just prior to the morning dose (trough sample).

When the randomized allocation requires a switch, the AED(s) currently taken (carbamazepine, valproic acid, topiramate, oxcarbazepine, levetiracetam and/or lamotrigine) will be substituted, starting with the morning dose on day 2, with an equivalent formulation available in the market. Namely, a brand product will be switched to a generic, randomly chosen among those available in the market, while maintaining unaltered the dosing regimen and times of administration.Likewise, a generic product will be switched to the brand or another generic, as determined by the randomization scheme, while maintaining unaltered the dosing regimen and times of administration. For AEDs which are commercially available both as immediate-release as well as sustained-release dose forms, the substituted product (brand of generic) will have equivalent release characteristics. The newly allocated treatments will be continued unchanged for 4 days (days 2,3,4 and 5) or 5 days (days 2,3,4, 5 and 6) for patients receiving lamotrigine or topiramate without enzyme inducers, or lamotrigine combined with enzyme inducers plus valproate. No changes in concomitant treatments will be allowed during the 5/6 days of the study, although addition, withdrawal or dose modification of drugs not interacting pharmacokinetically with the medications taken by the subject will be permitted.

When the randomized allocation requires continuation on the same product (control), the AED product(s) currently taken will be continued unaltered, with the same dosing regimen and times of administration. No changes in concomitant treatments will be allowed during the 5/6 days of the study, although addition, withdrawal or dose modification of drugs not interacting pharmacokinetically with the medications taken by the subject will be permitted.

In both the test and the control allocations, two further blood samples for the determination of the serum levels of the AED(s) will be collected again 4 days later (5 days later for patients remaining on randomized treatment for 5 days), one two hours after the evening dose (absorptive phase sample) on day 5 (day 6 for patients remaining on randomized treatment for 6 days) and one in the next morning (day 6 or 7) just prior to the morning dose (trough sample). Care will be taken to ensure that the samples on days 5 and 6/7 be collected at the same times, not only in relation to times of dosing but also in relation to actual time of the day and meal times. A 4-day interval for the post-randomization pharmacokinetic assessment is sufficient to reach steady state for AEDs with expected half-lives of about 12 h or less (carbamazepine, levetiracetam, valproic acid, topiramate combined with enzyme inducers, lamotrigine combined with enzyme inducers, and the monohydoxyderivative (MHD) of oxcarbazepine, for which oxcarbazepine is a prodrug). Likewise, a 5-day interval is sufficient to reach steady state for AEDs with expected half-lives of about 24 h (lamotrigine and topiramate not combined with enzyme inducers, and lamotrigine combined with both enzyme inducers and valproic acid).

All subjects will be kept under medical observation during the study with a daily unstructured interview and any additional investigation if needed, and any relevant change in clinical status, including any treatment-emergent adverse event, will be recorded in the CRF. During the 6/7-day observation period, subjects may undergo any clinical and laboratory investigations (eg., hematology and blood chemistry tests, neuroimaging tests, EEGs) as clinically indicated for their condition.

Patients will exit the study on day 6 or 7 as applicable and thereafter will be managed as considered indicated by the attending physician. This could involve substituting the AED product taken at that time in compliance with the policy on generic substitution implemented at that hospital.

If a change in dose of the AEDs being tested or any potentially interacting comedication is necessary prior to day 5/6, the two post-randomization samples may be collected 24 h earlier for AEDs with half lives of about 12 h or less (carbamazepine, levetiracetam, valproic acid, topiramate combined with enzyme inducers, MHD, and lamotrigine combined with enzyme inducers). Because in these patients the half-life of the AED being tested allows attainment of steady-steady conditions within 72 h. After collection of the post-randomization samples, the subject will exit the study. In all other situations requiring premature termination of the allocated treatment, subjects will exit the study and will be considered as drop-outs with no evaluable pharmacokinetic outcome data.

At enrollment (baseline), the subject's medical and pharmacological history and results of physical examination will be recorded. Historical data on seizure types and seizure frequency will be collected, and assessment of adverse effects of AED therapy by unstructured interview and application of the Adverse Event Profile (AEP) 21-item questionnaire developed by Baker et al. (1997) . The AEP questionnaire and the physical examination will be repeated on day 6/7. Occurrence of seizures will be recorded daily.

The AED products tested will include exclusively products commercially available in the Italian market. In accordance with the current regulation (DM 17.12.2012), the hospital pharmacy of each study site will stock the full range of available brand and generic products of study drugs sufficient to cover at least 6-day treatment at average dosages. All drug products will be stored, dispensed and tracked according to GCP guidelines.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older;
* currently being treated and at steady-state with any product (brand or generic) of carbamazepine, valproic acid, topiramate, oxcarbazepine, levetiracetam and/or lamotrigine administered in two or three divided daily doses, either alone or in combination with other drugs;
* a diagnosis of epilepsy or any other condition justifying prescription of AED therapy;
* being admitted to hospital (or being already in hospital) for observation/diagnostic evaluation or any other indication;
* expected to remain on the currently prescribed drug treatment for at least 5 days (or 6 days for patients receiving lamotrigine or topiramate without enzyme inducers, or receiving lamotrigine combined with enzyme inducers plus valproate);
* willingness to provide free, informed consent.

Exclusion Criteria:

* a history of known or suspected poor compliance;

  * recent changes in drug treatment, including potentially interacting comedication, which may have prevented attainment of steady-state conditions of the AED(s) being tested;
* known disorders of gastric motility;
* pregnancy or lactation;
* any condition which is expected to alter the pharmacokinetics of the study drug(s) over the subsequent 5/6 days;
* inability to fully understand the nature and implications of the study.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2012-05; Primary Completion 2015-05 (Estimated); Study Completion 2015-05 (Estimated)

PRIMARY OUTCOMES:
Serum drug concentration (25% change in serum drug concentration) | After six months
  The primary outcome endpoint will be the proportion of patients who post-randomization show a greater than 25% change in serum drug concentration compared with baseline. When comparing differences in serum concentration between post-randomization and baseline, the mean of the two values (post-absorptive and trough) measured on each occasion will be used because this provides a more accurate estimate of relative bioavailability.

SECONDARY OUTCOMES:
Serum drug concentration (15% change in mean serum drug concentration) | After six months
  proportion of patients who post-randomization will show a greater than 15% change in mean serum drug concentration compared with baseline
Serum drug concentration (50% change in mean serum drug concentration) | After six months
  proportion of patients who post-randomization will show a greater than 50% change in mean serum drug concentration compared with baseline
Serum drug concentration (5, 25% and 50% change in either post-absorptive or trough serum drug concentration) | After six months
  proportion of patients who will show a greater than 15, 25% and 50% change in either post-absorptive or trough serum drug concentration compared with baseline
Serum drug concentration (distribution in individual serum drug concentrations) | After six months
  distribution in individual serum drug concentrations post-randomization compared with baseline
Serum drug concentration (mean percent change (and %CV) in serum drug concentration) | After six months
  mean percent change (and %CV) in serum drug concentration post-randomization compared with baseline
adverse events | After three years
  proportion of patients with adverse events
adverse events | After three years
  adverse event (AEP) scores
first seizure after randomization | After three years
  interval elapsed between randomization and the first seizure
products (by type of AED, specific product utilized, and type of switch (brand to generic and generic to generic) | After three years
  the above outcome measures, by type of AED, specific product utilized, and type of switch (brand to generic and generic to generic).

CONTACTS AND LOCATIONS:
Overall Officials: Emilio Perucca, MD, Principal Investigator — IRCCS National Neurological Institute "C. Mondino" Foundation
Locations (16):
- Italy (16):
  - Clinica Neurologica Amaducci, Policlinico di Bari, Bari, Bari
  - Dipartimento di Scienze Neurologiche, Università degli Studi di Bologna, Bologna, Bologna
  - Azienda Ospedaliera, Policlinico Universitario Mater Domini, Catanzaro, Catanzaro
  - Azienda Ospedaliera ospedali Riuniti, Foggia, Foggia
  - Azienda Ospedaliera Universitaria Policlinico Gaetano Martino, Messina, Messina
  - UO di Neurologia, Azienda Ospedaliero Universitaria Pisana, Pisa, Pisa
  - Clinica Neurologica, Ospedali Riuniti, Ancona
  - U.S.C. Neurologia, Ospedali Riuniti, Bergamo
  - Unità Operativa Complessa di Neurologia, Ospedale di Bellaria, Bologna
  - Centro Regionale dell'Epilessia, Azienda Ospedaliera Spedali Civili, Brescia
  - Clinica Neurologica, Ospedale San Gerardo, Monza
  - Clinica Neurologica, Azienda Ospedaliero-Universitaria Maggiore della Carità, Novara
  - S.C. di Neurofisiopatologia, Centro di Riferimento Regionale Umbro per l'Epilessia, Perugia
  - Centro Regionale Epilessie, Reggio Calabria e Università della Magna Graecia, Reggio Calabria
  - Dipartimento di Scienze Neurologiche, III Clinica Neurologica, Università "La Sapienza", Roma
  - Unità Complessa di Neurologia, Ospedale SS. Giovanni e Paolo, Venezia

REFERENCES:
- [Background] Andermann F, Duh MS, Gosselin A, Paradis PE. Compulsory generic switching of antiepileptic drugs: high switchback rates to branded compounds compared with other drug classes. Epilepsia. 2007 Mar;48(3):464-9. doi: 10.1111/j.1528-1167.2007.01007.x. PMID 17346246
- [Background] Baker GA, Jacoby A, Buck D, Stalgis C, Monnet D. Quality of life of people with epilepsy: a European study. Epilepsia. 1997 Mar;38(3):353-62. doi: 10.1111/j.1528-1157.1997.tb01128.x. PMID 9070599
- [Background] Bartoli A, Marchiselli R, Gatti G. A rapid and specific assay for the determination of lamotrigine in human plasma by normal-phase HPLC. Ther Drug Monit. 1997 Feb;19(1):100-7. doi: 10.1097/00007691-199702000-00020. PMID 9029758
- [Background] Berg MJ, Gross RA, Tomaszewski KJ, Zingaro WM, Haskins LS. Generic substitution in the treatment of epilepsy: case evidence of breakthrough seizures. Neurology. 2008 Aug 12;71(7):525-30. doi: 10.1212/01.wnl.0000319958.37502.8e. PMID 18695164
- [Background] Berg MJ, Gross RA, Haskins LS, Zingaro WM, Tomaszewski KJ. Generic substitution in the treatment of epilepsy: patient and physician perceptions. Epilepsy Behav. 2008 Nov;13(4):693-9. doi: 10.1016/j.yebeh.2008.06.001. Epub 2008 Sep 10. PMID 18589000
- [Background] Bialer M, Midha KK. Generic products of antiepileptic drugs: a perspective on bioequivalence and interchangeability. Epilepsia. 2010 Jun;51(6):941-50. doi: 10.1111/j.1528-1167.2010.02573.x. Epub 2010 Apr 8. PMID 20384761
- [Background] Kramer G, Biraben A, Carreno M, Guekht A, de Haan GJ, Jedrzejczak J, Josephs D, van Rijckevorsel K, Zaccara G. Current approaches to the use of generic antiepileptic drugs. Epilepsy Behav. 2007 Aug;11(1):46-52. doi: 10.1016/j.yebeh.2007.03.014. Epub 2007 May 29. PMID 17537678
- [Background] Labiner DM, Paradis PE, Manjunath R, Duh MS, Lafeuille MH, Latremouille-Viau D, Lefebvre P, Helmers SL. Generic antiepileptic drugs and associated medical resource utilization in the United States. Neurology. 2010 May 18;74(20):1566-74. doi: 10.1212/WNL.0b013e3181df091b. Epub 2010 Apr 14. PMID 20393142
- [Background] Kesselheim AS, Stedman MR, Bubrick EJ, Gagne JJ, Misono AS, Lee JL, Brookhart MA, Avorn J, Shrank WH. Seizure outcomes following the use of generic versus brand-name antiepileptic drugs: a systematic review and meta-analysis. Drugs. 2010 Mar 26;70(5):605-21. doi: 10.2165/10898530-000000000-00000. PMID 20329806
- [Background] Perucca E, Albani F, Capovilla G, Bernardina BD, Michelucci R, Zaccara G. Recommendations of the Italian League against Epilepsy working group on generic products of antiepileptic drugs. Epilepsia. 2006;47 Suppl 5:16-20. doi: 10.1111/j.1528-1167.2006.00871.x. PMID 17239100
- [Background] Privitera MD. Generic antiepileptic drugs: current controversies and future directions. Epilepsy Curr. 2008 Sep-Oct;8(5):113-7. doi: 10.1111/j.1535-7511.2008.00261.x. PMID 18852829
- [Background] Zachry WM 3rd, Doan QD, Clewell JD, Smith BJ. Case-control analysis of ambulance, emergency room, or inpatient hospital events for epilepsy and antiepileptic drug formulation changes. Epilepsia. 2009 Mar;50(3):493-500. doi: 10.1111/j.1528-1167.2008.01703.x. Epub 2008 Jun 26. PMID 18616554
- [Background] Wilner AN. Therapeutic equivalency of generic antiepileptic drugs: results of a survey. Epilepsy Behav. 2004 Dec;5(6):995-8. doi: 10.1016/j.yebeh.2004.05.011. PMID 15582850